CLINICAL TRIAL: NCT03881020
Title: Comparison of Silver Modified and Conventional Atraumatic Restorative Treatment Modalities in Primary Molars in a Group of Egyptian School Children. A Randomized Controlled Trial
Brief Title: Comparison of Silver Modified and Conventional Atraumatic Restorative Treatment Modalities
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Abla Ahmed Mohamed Aly Ahmed, Assistant lecturer at Faculty of Oral and Dental Medicine Future University in Egypt, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PED 18-3D
Record Dates: First submitted 2019-03-11; First posted 2019-03-19 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SMART (Experimental): Silver modified atraumatic restorative treatment group in which advantage Arrest Silver diamine Fluoride 38% (Elevate oral Care, USA ) will be applied to carious molars then teeth will be restored with GC Fuji IX GP® FAST FAST Packable Posterior Restorative glass ionomer fillings (GC corporation, Tokyo, Japan)
  Interventions: Drug: Silver diamine Fluoride 38%
- Conventional ART (Active Comparator): Conventional atraumatic restorative treatment group in which a sharp excavator will be used to remove caries from carious molars then teeth will be restored with GC Fuji IX GP® FAST FAST Packable Posterior Restorative glass ionomer fillings (GC corporation, Tokyo, Japan)
  Interventions: Procedure: Conventional atraumatic restorative treatment

INTERVENTIONS:
Drug: Silver diamine Fluoride 38% — In the intervention group 38% Silver Diamine Fluoride will be applied to the surface of the isolated lesion for a period of 1 minute followed by glass ionomer restoration at the same visit.
  Other Names: Advantage Arrest Silver diamine Fluoride 38%
  Arms: SMART
Procedure: Conventional atraumatic restorative treatment — In the active comparator group caries will be removed from primary molars using sharp excavators then teeth will be restored using glass ionomer filling material at the same visit.
  Other Names: ART
  Arms: Conventional ART

SUMMARY:
The study is a randomized controlled trial aiming to compare the effectiveness of Silver modified atraumatic restorative technique and (SMART) and conventional atraumatic restorative technique (ART) regarding their caries arresting properties in primary molars, patient acceptance and cost effectiveness.

DETAILED DESCRIPTION:
5-9 years old school children will be recruited for the study. Parents of eligible children will be informed in full details about the purpose of the study and any possible side effects. Prior to enrollment of children in the study, parents will have to sign a written informed consent outlined by the Ethical Committee, Faculty of Dentistry, Ain Shams University. Children will be also informed about the nature of the study using age appropriate language and will have to give an assent to participate before being enrolled in the study.

Children will be clinically examined with the help of a plane dental mirror and an explorer. A single calibrated investigator will undertake all clinical examinations and deliver dental treatment to all patients to ensure standardization. After clinical examination, all children included in the study will be randomly allocated to be one of the two groups either control group (Conventional ART) or experimental group (SMART). Randomization sequence will be electronically generated using (http://randomization.com/). To ensure concealment of allocation, the randomly generated sequence will be concealed and enclosed in sealed, opaque envelopes. The envelopes will be randomly picked up by the children for group allocation. Follow up examinations will be done by a calibrated examiner who was not involved in the treatment procedures. Patients who are no longer willing to continue in the study will have the right to quit at any time without any penalty. All patient information will be collected and recorded in the patient examination chart. All information will be kept as a hard copy and as an electronic copy as well. Patient information will be confidential information that should never be exposed at any point. The data concerning the subjects will be entered into the database with a numerical code only for the purpose of confidentiality.

All data will be tabulated, summarized and statistically analyzed. Data will be statistically described in terms of mean, standard deviation, median and range, or frequencies (number of cases) and percentages when appropriate.

Comparison of numerical variables between the study groups will be done using Student t test for independent samples in comparing normally distributed data and Mann Whitney U test for independent samples when data is not normally distributed. For comparing categorical data, Chi-square test will be performed. Exact test will be used instead when the expected frequency is less than 5.Correlation between various variables will be done using Pearson moment correlation equation for linear relation in normally distributed variables and Spearman rank correlation equation for non-normal variables.

A probability value (p value) less than 0.05 is considered statistically significant. All statistical calculations will be done using computer programs Microsoft Excel 2007 (Microsoft Corporation, NY, USA) and IBM SPSS (Statistical Package for the Social Science; IBM Corp, Armonk, NY, USA) release 22 for Microsoft Windows.

ELIGIBILITY:
Inclusion Criteria:

1. Medically free children.
2. Clinical examination revealing at least one second primary molar with single surface active dentine carious lesions.
3. Children who agreed to participate and whose parents signed an informed consent.
4. Cooperative or potentially cooperative children according to Wright Classification

Exclusion Criteria:

1. Children who have known allergies to silver products.
2. Children with special health care needs or any medical conditions.
3. Children with designated molars having more than one third of their crown missing.
4. Children with designated molars showing signs of pulpal pathology such as spontaneous pain, presence of an abscess or sinus or mobility.
5. Children with designated molars having an existing restoration.
6. Children with designated molars having deep carious lesions with close proximity to the pulp.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Arresting carious lesion progression and restoration survival | 1 year
  Restorations will be assessed for clinical success and caries arrest in terms of presence of sensitivity, marginal integrity, restoration survival and recurrent caries using United States Public Health Services (USPHS) criteria. Restorations with good color match, good marginal adaptation, no sensitivity and no evidence of caries will be given score alfa (A).
  Restorations with slight discoloration, slight discontinuity and diminishing sensitivity will be given score bravo (B). Restorations with unacceptable color, exposed dentin, constant sensitivity and evidence of caries will be given score charlie (C). Restorations fractured or lost will be scored as delta (D).

SECONDARY OUTCOMES:
Patient acceptance | will be recorded immediately after the procedure
  Patient acceptance will be recorded by using self-reported approach to assess the level of child discomfort using the Wong-Baker Facial Scale. The scale shows a series of faces ranging from a happy face to a crying face. The patients will choose the face that best describes their level of pain. The first face represents a pain score of 0 which indicates "no hurt". The second face represents a pain score of 2 which indicates "hurts a little bit." The third face represents a pain score of 4, which indicates "hurts a little more". The fourth face represents a pain score of 6 which indicates "hurts even more". The fifth face represents a pain score of 8 which indicates "hurts a whole lot"; the sixth face represents a pain score of 10 indicating "hurts worst".

OTHER OUTCOMES:
cost effectiveness | 1 year
  The average cost per restoration will be calculated for both treatment modalities, whereas the effectiveness will be estimated in terms of restoration survival over the 1 year follow up. Cost effectiveness will be calculated by dividing the average cost per restoration by the survival of the restoration after 1 year .

CONTACTS AND LOCATIONS:
Overall Officials: Abla Ah Aly, A. Lecturer, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aly AAM, Aziz AMA, Elghazawy RK, El Fadl RKA. Survival Analysis and Cost Effectiveness of Silver Modified Atraumatic Restorative Treatment (SMART) and ART Occlusal Restorations in Primary Molars: a randomized controlled trial. J Dent. 2023 Jan;128:104379. doi: 10.1016/j.jdent.2022.104379. Epub 2022 Nov 29. PMID 36460236